CLINICAL TRIAL: NCT03458897
Title: Quantitative MRI for Patients With Sickle Cell Disease Undergoing Hematopoietic Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ghada Abusin, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00132776
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Sickle Cell Disease
Keywords: bone marrow cellularity; bone marrow transplant
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI arm (Experimental): Subjects with sickle cell disease undergoing bone marrow transplantation will undergo serial functional MRI (up to 4 scans).
  Interventions: Diagnostic Test: serial functional magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: serial functional magnetic resonance imaging (MRI) — All subjects with sickle cell disease undergoing bone marrow transplantation will undergo up to 4 functional MRI scans.

SUMMARY:
The primary purpose of this research is to determine if it is feasible to perform serial magnetic resonance imaging (MRI) to evaluate the amount of bone marrow cells (also called cellularity) and iron stores before and after bone marrow transplantation for severe sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years.
* Diagnosis of SCD ([Hemoglobin SS (Hb-SS), Hemoglobin SC (Hb-SC) or Hemoglobin S-Beta thalassemia (Hb-Sβ) genotype].
* Patient is a candidate for an allogeneic HCT.
* Subject or guardians have given informed consent.

Exclusion Criteria

* The need for general anesthesia for MRI.
* Subjects with implanted magnetic devices (e.g. pacemakers) that may malfunction or move in the strong magnetic field.
* A subject who is pregnant.
* Previous HCT.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of obtaining serial scans in patients with sickle cell undergoing marrow transplant | 110 days post transplant
  Feasibility will be measured by the number of subjects who undergo at least 2 of 4 scheduled functional MRI's

SECONDARY OUTCOMES:
MRI and hemoglobin S. | 1 year post transplant
  Correlation between functional MRI result and hemoglobin S level.
MRI and neutrophil engraftment | 1 year post transplant
  Correlation between functional MRI result and time to neutrophil engraftment
MRI and chimerism | 1 year post transplant
  Correlation between functional MRI result and time to donor/ recipient chimerism

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abusin, MBBS MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No